CLINICAL TRIAL: NCT02346032
Title: Phase II Study of Refametinib, a MEK Inhibitor, as Second-line Treatment in Advanced Biliary Tract Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ho Yeong Lim, MD, Ph.D, Devision of hematology-oncology, Department of medicine, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-07-148
Record Dates: First submitted 2014-11-18; First posted 2015-01-26 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Biliary Tract Cancer
Keywords: second line
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — N-(3,4-difluoro-2-(2-fluoro-4-iodophenylamino)-6-methoxyphenyl)-1-(2,3-dihydroxypropyl)cyclopropane-1-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- refametinib (Experimental): refametinib medication
  Interventions: Drug: refametinib

INTERVENTIONS:
Drug: refametinib — Refametinib will be administered orally at the starting dose of 50 mg twice daily on a continuous daily dosing schedule.

SUMMARY:
Phase II Study of Refametinib, a MEK inhibitor, as second-line treatment in advanced biliary tract adenocarcinoma

DETAILED DESCRIPTION:
Refametinib will be administered orally at the starting dose of 50 mg twice daily on a continuous daily dosing schedule.

Self-administration of refametinib tablets will take place on an outpatient basis. Patients experiencing dose-limiting toxicity attributed to study medication should have at least 1-week treatment breaks inserted into the continuous daily dosing period as needed and/or may be interrupted or reduced depending on individual tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18
2. histologically or cytologically confirmed adenocarcinoma of biliary tract
3. unresectable or metastatic
4. ECOG performance status of 0~2
5. measurable lesion per RECIST 1.1 criteria
6. adequate marrow, hepatic, renal functions
7. normal range of cardiac function confirmed by echocardiogram within 1 year (LVEF ≥50)
8. Child-Pugh Class A in case of liver cirrhosis
9. One prior treatment of cytotoxic chemotherapy (including adjuvant treatment within 12 months)
10. Resolution of all acute toxic effects of any prior therapy to Common Toxicity Criteria for Adverse Events (CTCAE 4.03) ≤ grade 1.
11. provision of a signed written informed consent

Exclusion Criteria:

1. History of cardiac disease
2. Ongoing infection > Grade 2 according to NCI-CTCAE version 4.03. Hepatitis B is allowed if no active replication (defined as abnormal ALT >2xULN associated with HBV DNA >20,000 IU/mL) is present
3. Severe co-morbid illness and/or active infections including active hepatitis C and human immunodeficiency virus (HIV) infection
4. History of interstitial lung disease (ILD).
5. Any cancer curatively treated < 3 years prior to study entry, except cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors (Staging: Ta, Tis and T1).
6. Renal failure requiring hemo- or peritoneal dialysis.
7. Clinically significant GI bleeding (CTCAE 4.03 grade 3 or higher) within 30 days prior to start of screening
8. Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks) within 6 months prior to start of screening.
9. History of organ allograft, cornea transplantation will be allowed
10. Active CNS metastases not controllable with radiotherapy or corticosteroids
11. Visible retinal pathology as assessed by ophthalmologic exam that is considered a risk factor for RVO or CSR.
12. Known history of hypersensitivity to study drugs
13. Any condition that was unstable or which could jeopardize the safety of the patient and his/her compliance in the study
14. Non-healing wound, ulcer, or bone fracture.
15. Patients with seizure disorder requiring medication.
16. Use of strong inhibitors of CYP3A4 and strong inducers of CYP3A4 should be stopped 2 weeks before start of screening (see Appendix 1).
17. Acute steroid therapy or taper for any purpose (chronic steroid therapy is acceptable provided that the dose is stable for 1 month before start of screening and thereafter).
18. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
19. Pregnant or lactating women. Women of childbearing potential not employing adequate contraception. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to start of study treatment and a negative result must be documented before first dose of study drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-10-13 (Actual)

PRIMARY OUTCOMES:
Response rate | 12months
  the rate of complete response and partial response among all evaluable patients

SECONDARY OUTCOMES:
adverse events in each cycle were documented based on CTCAE v 4.03 | 24months
Duration of response | 12months
  median time from response to progression
Progression-free survival | 6months
Exploratory correlative analysis | 15 days
  KRAS/PIK3CA mutation testing using BEAMing assay will be planned
Overall survival | 12months